CLINICAL TRIAL: NCT01216228
Title: Food Patterns, Inflammation Markers of Cardiovascular Disease Risk and Incidence of CVD
Status: Completed | Type: Observational
Sponsor: Skane University Hospital (Other)
Responsible Party: Jan Nilsson, Professor, Lund University
Other Study IDs: MKC 2010-10-06
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Last update posted 2010-10-07 (Estimated); Status verified 2006-10

CONDITIONS: Cardiovascular Disease; Diet; Inflammation
MeSH Terms: conditions — Cardiovascular Diseases; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Health outcome studies should examine food patterns, because foods are consumed together and nutrients are metabolized jointly. To examine associations between food patterns and markers of systemic and vascular inflammation at baseline, in a population-based cohort in Malmö, Sweden, and after 13 years of follow-up food pattern associations with CVD incidence.

ELIGIBILITY:
Inclusion Criteria:

* The "cardiovascular sub-cohort" is a random sample (i.e., 50 percent) of those who joined from November 1991 to February 1994. This group underwent additional examinations to assess carotid arteriosclerosis by ultrasound (n = 6103) and donated blood after fasting (n = 5533).

Exclusion Criteria:

* Subjects were excluded, either because they were using medication for diabetes mellitus or had previously been diagnosed as having diabetes mellitus.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The Malmö Diet and Cancer Cohort (MDC), a large-scale, population-based, prospective cohort study, was designed in the early 1990s to identify dietary and lifestyle risk factors related to the incidence of cancer. Men aged 46-73 years (n =11 063) and women aged 45-73 years (n = 17 035) living in Malmö, the third largest city in Sweden, at that time, were examinedinvited to participate. Baseline examinations took place at the MDC CentreCenter at the Skåne Malmö University Hospital in Malmö between March 1991 and October 1996.
Sampling Method: Non-Probability Sample
Dates: Start 1991-03